CLINICAL TRIAL: NCT06755398
Title: The Effect of Cognitive-Based Neuromuscular Exercises on Reaction Time, Joint Position Sense, Proprioceptive Force Sense and Balance in Individuals Who Had Anterior Cruciate Ligament Surgery
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ertuğrul Demirdel (Other)
Collaborators: Antalya Bilim University (Other)
Responsible Party: Sponsor-Investigator, Ertuğrul Demirdel, Associate professor, Ankara Yildirim Beyazıt University
Organization: Ankara Yildirim Beyazıt University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AnkaraYBU-OA
Record Dates: First submitted 2024-12-18; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-06

CONDITIONS: ACL - Anterior Cruciate Ligament Rupture
Keywords: ACL rupture; Cocnitive task; Proprioception; Dual Task
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard treatment group (Sham Comparator): The protocol developed by the Royal Dutch Society for Physical Therapy (KNGF) will be applied following anterior cruciate ligament (ACL) surgery.
  Interventions: Other: Exercise
- experimental group (Experimental): During the exercises based on the protocol developed by the Royal Dutch Society for Physical Therapy (KNGF) following anterior cruciate ligament (ACL) surgery, additional cognitive tasks will be assigned to the patients.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — During the exercises based on the protocol developed by the Royal Dutch Society for Physical Therapy (KNGF) following anterior cruciate ligament (ACL) surgery, additional cognitive tasks will be assigned to the patients.
  Other Names: dual task exercises; cognitive exercises
  Arms: Standard treatment group
Other: Exercise — The protocol developed by the Royal Dutch Society for Physical Therapy (KNGF) will be applied following anterior cruciate ligament (ACL) surgery.
  Other Names: exercises
  Arms: experimental group

SUMMARY:
The aim of this study is to investigate the effects of cognitive-based neuromuscular exercises on increased reaction time, decreased joint position sense, reduced proprioceptive force sense, and balance problems in individuals who have undergone surgery following anterior cruciate ligament (ACL) injuries. With the results obtained from the study, the investigators aim to provide a different perspective on rehabilitation methods applied after ACL reconstruction and contribute to the literature with objective and evidence-based information regarding the effects of cognitive-based neuromuscular exercises on sensorimotor, neuromuscular, and proprioceptive senses.

DETAILED DESCRIPTION:
Anterior Cruciate Ligament (ACL) injuries are among the most common knee injuries, occurring due to both contact and non-contact mechanisms, such as sudden deceleration, changes in direction, or landing after jumping, and leading to disruptions in knee stability and biomechanics. In the United States, it is estimated that there are between 100,000 and 200,000 cases annually, while the global incidence of ACL ruptures approaches 2 million cases per year. Treatment for ACL injuries can be either conservative or surgical. Conservative treatment is considered a viable option for specific populations, such as athletes who do not engage in activities requiring direction changes, individuals with no significant knee instability, and those with lower activity levels. ACL injuries result in quadriceps and hamstring weakness, reduced knee joint proprioception, and impaired balance.

To restore the anatomy and biomechanics of the knee, arthroscopic ACL reconstruction is performed to stabilize the knee and prevent secondary injuries, with approximately 30,000 procedures conducted annually in the United Kingdom. Although comprehensive rehabilitation is a critical component of ACL injury management, whether treated conservatively or surgically, there is currently no gold standard rehabilitation approach for such a widespread injury.

The type of rehabilitation protocol applied is one of the most significant factors influencing the outcomes of ACL reconstruction. Rehabilitation protocols have evolved substantially over the past few decades, with traditional rehabilitation, accelerated rehabilitation, and criterion-based rehabilitation protocols being the most commonly employed. These protocols aim to enhance muscle strength, improve proprioception, and ensure knee stabilization, with the timing and types of exercises determined by the biological healing and remodeling periods of the graft.

Criterion-based rehabilitation protocols, a relatively new approach, aim to provide patient-specific rehabilitation and maximize progress. Developed in 2016 by the Royal Dutch Society for Physical Therapy (KNGF), this protocol is divided into three phases: early, mid, and late stages. To progress to the next stage, patients must meet specific goals for each phase, which are verified through objective and subjective testing. The effectiveness and quality of early and mid-stage rehabilitation significantly influence long-term outcomes. The goals of early-stage rehabilitation, lasting approximately two months, include reducing effusion, restoring joint range of motion, and minimizing muscle atrophy. During the mid-stage, which extends from the second to the sixth month, the focus shifts to achieving full control of knee extension, restoring 80% of the muscle strength in the operated limb compared to the uninjured side, and regaining jumping ability. This phase includes exercises such as knee flexor and extensor strengthening, closed kinetic chain exercises, functional exercises, balance training, plyometric exercises, and neuromuscular exercises.

Neuromuscular control is essential for initiating movement and requires the integration of sensory information from proprioceptive, kinesthetic, visual, and vestibular sources, as well as cortical and spinal motor commands. This control is critical for the effective execution of movement. Recent studies indicate that ACL injuries are not isolated joint damages that merely affect stability and biomechanics but also directly influence neuromuscular control of the knee via mechanoreceptors located within the ACL. These injuries lead to neurophysiological effects on sensorimotor control. Following ACL injuries, these somatosensory changes may result in deficits in postural and motor control, leading to slower lower extremity reaction times. Additionally, nociceptive activity related to pain and swelling, combined with reduced joint position sense and kinesthesia, impairs movement quality. Neuromuscular control impairments, proprioceptive deficits, and disruptions in somatosensory inputs due to damaged mechanoreceptors may persist for 9-12 months, highlighting the need for targeted exercises during the mid-stage rehabilitation.

The complex integration of vestibular, visual, and somatosensory inputs, necessary for situational awareness, enhanced alertness, and the ability to select between attentional resources, can promote the development of neurocognitive functions. Cognitive-based neuromuscular exercises aim to improve patients' reaction times, joint position sense, proprioceptive strength, and neurocognitive functions such as balance, while enhancing motor control and knee stability. An example of cognitive-based neuromuscular exercises is the Life Kinetik (LK) method, developed by Lutz in Germany in 2007. This method is used to promote neural learning, support neuroplasticity, and reduce neurological symptoms. During these exercises, visual or cognitive tasks are combined with physical activity to train the brain, aiming to enhance concentration, problem-solving skills, reflexes, balance, and coordination. These exercises involve performing multiple complex tasks that require active and continuous thinking during movements. The investigators hypothesize that the complex tasks involved in these exercises may positively influence reaction time, joint position sense, proprioceptive strength, and balance, which are impaired following ACL reconstruction.

A review of the literature reveals that studies examining joint position sense, neurocognitive control, and reaction time in patients undergoing ACL reconstruction are limited. Furthermore, research investigating lower extremity reaction or detection time, resulting from disrupted somatosensory inputs after ACL injuries, is also scarce. While studies have been conducted on neuromuscular exercises in ACL rehabilitation programs, no research has been identified focusing on cognitive-based neuromuscular exercises. The lack of a gold standard rehabilitation method for ACL reconstruction in the literature has driven ongoing research into new treatment modalities and their effects. Recently, cognitive-based neuromuscular exercises have emerged as a promising method to enhance cognitive abilities, joint position sense, perceptual strength, and balance.

This study is designed to investigate the effects of cognitive-based neuromuscular exercises on reaction time, joint position sense, proprioceptive force sense, and balance disorders observed in patients following anterior cruciate ligament (ACL) reconstruction. With the results obtained from this study, the investigators aim to provide a new perspective on rehabilitation approaches in ACL reconstruction, where no gold standard treatment exists, and contribute to the literature with objective and evidence-based data regarding the effects of cognitive-based neuromuscular exercises on sensorimotor, neuromuscular, and proprioceptive senses.

Study Population and Sample The study will include individuals of both genders aged 20-40 years. Post-surgical patients will initially undergo an 8-week home-based rehabilitation program, as described by McNeil et al., with weekly monitoring to assess their progress. At the end of the 8th week, patients who meet the criteria for the early phase of a criterion-based rehabilitation approach will be included in the study. These participants will then follow an 8-week rehabilitation program, twice per week, adhering to the mid-phase criterion-based rehabilitation protocol. All rehabilitation sessions will be conducted in-person under the supervision of an experienced physiotherapist. Measurements will be performed before the rehabilitation and at the end of the 8-week program. The sample size was calculated using G*Power 3.1, and a total of 27 participants were determined with 80% power.

Data Collection Tools Demographic data, including age, gender, body weight, height, BMI, alcohol and smoking habits, injured limb, time between injury and surgery, and occupation, will be collected.

Pain Measurement: Pain intensity will be assessed using the Numeric Pain Scale (0 = no pain, 10 = worst imaginable pain).

Lower Extremity Reaction Time Measurement: FITLIGHT Corp, a wireless light-sensor system, will be used to measure reaction time. Participants will deactivate randomly lit sensors using the affected and unaffected lower extremities. Task variations will include cognitive dual tasks (e.g., counting backward by fives) and motor dual tasks (e.g., tossing and catching a ball) to assess dual-task performance.

Joint Position Sense: Passive joint position sense will be evaluated using a joint repositioning task at 15° and 45° knee flexion, with measurements taken using the "Clinometer" smartphone application. Cognitive and motor tasks will also be incorporated.

Proprioceptive Force Sense: Proprioceptive force sense will be assessed using the StabilizerTM biofeedback device. Participants will perform isometric contractions, and differences between targeted and actual force values will be recorded. Cognitive and motor dual tasks will also be included.

Static Balance Test: Single-leg stance tests will evaluate static balance under open-eye conditions. Dual-task conditions will include verbal tasks (e.g., naming words starting with specific letters) and motor tasks (e.g., holding a tray with a cup of water).

Activity Level: Pre-injury activity levels will be measured using the Tegner Activity Scale, which scores activity from 0 (no activity) to 10 (elite-level competition).

IKDC Subjective Knee Form: Knee symptoms, function, and activity levels will be evaluated using the International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Form. The total score ranges from 0 to 100, with higher scores indicating better function.

Treatment Protocol

Participants meeting progression criteria will undergo an 8-week mid-phase rehabilitation program (twice weekly). Patients will be randomly assigned to two groups:

Group 1: Exercises performed without secondary tasks. Group 2: Exercises performed with cognitive or motor dual tasks (e.g., rhythmic counting, reverse spelling, ball manipulation).

Example Exercises (Weeks 8-16):

Quadriceps and hamstring strengthening exercises, Hip, lumbo-pelvic, and gastrocnemius-soleus strengthening, Closed kinetic chain exercises, Functional exercises (e.g., squats, lunges, leg press), Balance training (e.g., tandem walking, single-leg stance with open and closed eyes).

Exercises will include 8-12 repetitions across 3 sets, ensuring optimal loading without over-stressing healing tissues. Pain and swelling will be closely monitored, with exercise intensity adjusted as necessary. Resistance will start at 40-50% of the unaffected limb's capacity and progress to 70-80%, depending on the patient's functional status.

ELIGIBILITY:
Inclusion Criteria:

* Having sustained a unilateral isolated anterior cruciate ligament injury,
* Having undergone anterior cruciate ligament reconstruction using a hamstring graft by a surgeon at least 8 weeks ago,
* Having completed the early phase of the postoperative criterion-based rehabilitation protocol and met the criteria for progression to the intermediate phase of the rehabilitation program (1- pain between 0-2 on the numeric pain scale, 2- no effusion in the knee, 3- no limitation in passive knee extension, 4- passive knee flexion of at least 120°, 5- full quadriceps activation (patient able to perform 10 repetitions of a single-leg raise exercise), and 6- normalized gait pattern without assistance).

Exclusion Criteria:

* Having a partial ACL tear,
* Having sustained bilateral ACL injuries,
* Having additional injuries accompanying the ACL injury,
* Having undergone ACL revision surgery,
* Having a history of complex knee surgery,
* Having any neurological, orthopedic, or systemic disease that may contraindicate exercise.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The Effect of an 8-Week Cognitive-Based Neuromuscular Exercise Program on Lower Extremity Reaction Time | 8 week
  This study evaluates lower extremity reaction time in individuals with anterior cruciate ligament (ACL) injuries using the FITLIGHT Corp system. Participants will deactivate randomly illuminated lights with their lower extremities. The system's wireless sensor discs will be placed according to each participant's leg length to minimize balance-related factors. Five lights will be arranged in a semicircular pattern at 45-degree intervals.
  Reaction time will be measured under three conditions: baseline, cognitive task, and motor task. In the baseline condition, participants will complete a 30-second practice trial followed by a 1-minute test trial. During the cognitive task, participants will count backward from 600 by fives while deactivating the lights. In the motor task, they will toss and catch a ball with their dominant hand while performing the light-deactivation task. The average reaction time in seconds will be recorded for both the injured and uninjured limbs.

CONTACTS AND LOCATIONS:
Overall Officials: Ertugrul Demirdel, Associate professor, Study Director — Ankara Yildirim Beyazıt University
Locations (1):
- Antalya Bilim University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Under the Personal Data Protection Law, disclosing personal data outside of official authorities constitutes a criminal offense. Additionally, the results of the study do not involve personal information.

REFERENCES:
- [Background] Elabd OM, Elabd AM. Functional outcomes of a criterion-based rehabilitation protocol for anterior cruciate ligament reconstruction in amateur athletes: A randomised clinical trial. J Bodyw Mov Ther. 2023 Jul;35:7-13. doi: 10.1016/j.jbmt.2023.04.037. Epub 2023 Apr 17. PMID 37330806
- [Background] Buckthorpe M, Della Villa F. Optimising the 'Mid-Stage' Training and Testing Process After ACL Reconstruction. Sports Med. 2020 Apr;50(4):657-678. doi: 10.1007/s40279-019-01222-6. PMID 31782065
- [Background] Elabd OM, Alghadir AH, Ibrahim AR, Hasan S, Rizvi MR, Sharma A, Iqbal A, Elabd AM. Functional outcomes of accelerated rehabilitation protocol for anterior cruciate ligament reconstruction in amateur athletes: a randomized clinical trial. J Rehabil Med. 2024 Feb 22;56:jrm12296. doi: 10.2340/jrm.v56.12296. PMID 38385715
- [Background] Li D, Zhang Q, Liu X, Chen C, Lu J, Ye D, Li Y, Wang W, Shen M. Effect of water-based walking exercise on rehabilitation of patients following ACL reconstruction: a prospective, randomised, single-blind clinical trial. Physiotherapy. 2022 Jun;115:18-26. doi: 10.1016/j.physio.2021.11.003. Epub 2021 Dec 1. PMID 35101723
- [Background] Kiele D, Solianik R. Four-Week Application of Kinesiotaping Improves Proprioception, Strength, and Balance in Individuals With Complete Anterior Cruciate Ligament Rupture. J Strength Cond Res. 2023 Jan 1;37(1):213-219. doi: 10.1519/JSC.0000000000004245. Epub 2022 Apr 13. PMID 35438677
- [Background] Buckthorpe M, Gokeler A, Herrington L, Hughes M, Grassi A, Wadey R, Patterson S, Compagnin A, La Rosa G, Della Villa F. Optimising the Early-Stage Rehabilitation Process Post-ACL Reconstruction. Sports Med. 2024 Jan;54(1):49-72. doi: 10.1007/s40279-023-01934-w. Epub 2023 Oct 3. PMID 37787846
- [Background] Leal J, Mirza B, Davies L, Fletcher H, Stokes J, Cook JA, Price A, Beard DJ. Cost-effectiveness analysis of a pragmatic randomized trial evaluating surgical reconstruction versus rehabilitation in patients with long-standing anterior cruciate ligament injury. Bone Joint J. 2024 Jan 1;106-B(1):38-45. doi: 10.1302/0301-620X.106B1.BJJ-2023-0175.R1. PMID 38160685